CLINICAL TRIAL: NCT04764240
Title: Prognostic Value of Examined and Metastatic Lymph Nodes in Chinese Esophageal Squamous Cell Carcinoma Patients Received Lymphadenectomy
Brief Title: Precisely Estimation of the Prognostic Value of Lymph Node in ESCC
Status: Completed | Type: Observational
Sponsor: Shanghai Cancer Hospital, China (Other)
Responsible Party: Sponsor
Other Study IDs: ASJSTO1901
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Lymph Node Excision

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: R0 resection with lymphadenectomy — Patients received a surgical R0 resection; patients who received an R1 or R2 resection were excluded.

SUMMARY:
Data were collected on a large multi-institution dataset consisting of ESCC patients who underwent surgery between January 2003 and December 2013 at ten institutions in the People's Republic of China. The datasets were approved for research by the institutional review board of each participating center. Prior to surgery, all patients received computerised tomography (CT) of the chest and abdomen and EUS as part of their routine staging workup. Patients received whole body FDG-PET to eliminate the possibility of distant metastases if the attending physician considered it was necessary. All patients in the dataset received a surgical R0 resection; patients who received an R1 or R2 resection were excluded. Notably, there is nothing approaching a consensus on the extent of lymph node dissection for ESCC patients. Patients who received neoadjuvant therapy were excluded due to the influence of neoadjuvant therapy on lymph node status and pathologic T stage. The primary endpoints were overall survival (OS), which was defined as the time between surgical resection and death from any cause, and cancer-specific survival (CSS), defined as the time from surgical resection to death caused by ESCC. After receiving esophagectomy, patients were followed up by clinical examination every three months for the first year, every three to six months for the second year, and every six to twelve months from then on.

ELIGIBILITY:
Inclusion Criteria:

1. Minimum age: 18 years
2. Patients underwent R0 resection and lymphadenectomy.
3. ECOG PS less than or equal 2
4. Adequate bone marrow function: Leukocytes > 3,5 x 10^9/L Absolute neutrophil count > 1,5 x 10^9/L Platelet count > 100 x 10^9/L Hemoglobin > 10 g/dl
5. Adequate hepatic function: Total bilirubin < 2,0 mg/dl ALAT, ASAT, alkaline phosphatase, gamma-GT < 3 x ULN 7. Serum creatinine < 1,5 mg/dl, creatinine-clearance > 50 ml/min
6. Written informed consent before randomization

Exclusion Criteria:

1. R1 or R2 resection
2. Patients underwent neoadjuvant therapy
3. Fertile patients without adequate contraception during therapy
4. Psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
5. History of severe somatic or psychological diseases: - instable cardiac disease not well controlled with medication, myocardial infarction within the last 6 months:* Central nervous system disorders or psychiatric disability including dementia or epileptic disease; * active uncontrolled intercurrent infections or sepsis
6. Previous or concurrent malignancies, with the exception of adequately treated basal cell carcinoma of the skin or in situ carcinoma of the cervix. The inclusion of patients with other adequately treated tumors within the last 5 years has to be discussed with the principal investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients elder than 18 years old received computerised tomography (CT) of the chest and abdomen and EUS as part of their routine staging workup. Patients received whole body FDG-PET to eliminate the possibility of distant metastases if the attending physician considered it was necessary. Patients underwent R0 resection and lymphadenectomy.
Sampling Method: Probability Sample
Enrollment: 3700 (Actual)
Dates: Start 2003-01-01 (Actual); Primary Completion 2013-12-30 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
OS | Five years
  Overall survival

IPD SHARING:
Plan to Share IPD: No